CLINICAL TRIAL: NCT01504620
Title: Performance Evaluation of BGStar and iBGStar in Terms of Accuracy (Polaris), Intra-assay Precision, and Hematocrit Interference (Helios Substudy) Following ISO15197 and TNO Guidelines
Brief Title: Performance Evaluation of Blood Glucose Monitoring Systems
Acronym: Polaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IKFE Institute for Clinical Research and Development (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BGSTA_C_05445; SAN-HCT-002 Helios (Other: IKFE); SAN-BGM-002 Precision (Other: IKFE)
Record Dates: First submitted 2011-12-27; First posted 2012-01-05 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; blood glucose self-assessment; Accuracy; Intra-Assay precision; Hematocrit interference
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar infusion (Other): Diagnostic assessment of blood glucose by means of different devices
  Interventions: Other: Sugar infusion
- insulin infusion (Experimental): infusion of insulin to achieve low glucose levels
  Interventions: Drug: insulin infusion

INTERVENTIONS:
Other: Sugar infusion — Infusion of glucose to achieve high blood glucose levels
  Other Names: 5 % glucose solution
  Arms: Sugar infusion
Drug: insulin infusion — i.v. infusion of insulin
  Other Names: insuman rapid
  Arms: insulin infusion

SUMMARY:
The goal of this single-center, comparative, open label, in-vitro diagnostic device performance evaluation was to investigate the performance of two sanofi-aventis BGMSs (BGStar® and iBGStar®) with regard to system accuracy (Polaris), precision and Hct influence (Helios).

DETAILED DESCRIPTION:
The main study (Polaris) investigated blood glucose measuring accuracy and intra-assay precision while the substudy (Helios) investigated potential haematocrit interference of sanofi-aventis BGMSs BGStar® and iBGStar® and partly of competitor BGMSs according to ISO 15197 [1] and TNO 2001 Quality Guideline [2], respectively.

The primary objective of the system accuracy evaluation is to identify the number of blood glucose readings of both sanofi-aventis devices within the ISO 15197 area of acceptable accuracy of ± 20% [DEV%] for blood samples with glucose concentration > 75 mg/dL (4.2 mmol/L) and within the ISO 15197 area of acceptable accuracy of ± 15 mg/dL (± 0.83 mmol/L) for blood samples with glucose concentration < 75 mg/dL (4.2 mmol/L) as compared to the StatStrip® Connectivity reference method. The primary objective of the haematocrit interference evaluation is to demonstrate that the BGStar® and iBGStar® devices meet the Hct interference requirements according to TNO 2001 Quality Guideline when used to measure BG of venous whole blood as compared to a venous plasma reference method (YSI 2300 STAT Plus™) at Hct levels between 35 - 55% in terms of:(1) a mean deviation not exceeding ± 10% [DEV%] for hyperglycaemic glucose concentrations (150 - 180, 250 - 280, 320 - 350 mg/dL) and (2)a mean deviation not exceeding ± 18 mg/dL (1.0 mmol/L) [DEVtotal] for hypo- and normoglycaemic glucose values (50 - 60, 100 - 120 mg/dL) compared to the reference method at Hct levels between 35 - 55%.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects or patients with type 1 or type 2 diabetes
* screening glucose levels fall into required glucose ranges
* screening hematocrit values between 36 % to 55 %

Exclusion Criteria:

* history of hypotension during blood draws
* intake of drugs known to interfere with blood glucose readings
* biochemical safety parameters outside of reference ranges
* Hb < 11 g/dL
* lack of compliance
* history of frequent hypoglycemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of the blood glucose meter in comparison to a standard reference | within 10 min up to 300 min after start of experiment
  After start of the experiment, blood glucose will be measured by means of the test devices and blood will be drawn for assessment of venous blood glucose concentration with a standard laboratory reference method

SECONDARY OUTCOMES:
Intra-Assay precision | within 10 min up to 300 min after start of experiment
  Blood samples from 5 individuals with different levels of blood glucose were each measured with 10 meters of both investigational devices, the BGStar® and iBGStar®, ten times resulting in a total number of 500 measurements.
Hematocrit Interference (Helios) | within 10 min up to 300 min after start of the experiment
  One patient provided blood and artificial samples are generated from venous heparinized blood. These blood samples were adjusted to five different BG levels (2.8 mmol/L, 5.6 mmol/L, 8.3 mmol/L, 13.9 mmol/L, 19.4 mmol/L) at five different Hct levels (35%, 40%, 45%, 50%, 55%) to fulfill the range required by the TNO 2001 and tested by all devices.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pfützner, MD, PhD, Principal Investigator — IKFE Institute for Clinical Research and Development
Locations (1):
- IKFE - Institute for Clinical Research and Development, Mainz, Germany